CLINICAL TRIAL: NCT01892956
Title: Observational Study of Blood Glucose Levels and Gut Microbiota in Healthy Individuals
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Other Study IDs: TASMC-12-ZH-658
Record Dates: First submitted 2013-05-26; First posted 2013-07-08 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Nutritional and Metabolic Diseases; Endocrine System Diseases; Disorders of Environmental Origin
MeSH Terms: conditions — Nutritional and Metabolic Diseases; Endocrine System Diseases; Disorders of Environmental Origin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood count, lipids, liver functions, CBP Stool sample for intestinal microbiota
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy volunteers
- Newly diagnosed T2DM: Newly diagnosed T2DM, who have not started yet medical treatment with glucose lowering medications
  Interventions: Other: Nutritional intervention

INTERVENTIONS:
Other: Nutritional intervention — 2 dietary interventions
  1. personalized diet based on algorithm predictions of glucose response to foods
  2. Mediterranean-style diet
  Groups: Newly diagnosed T2DM

SUMMARY:
Categorization of glucose levels into 'healthy', 'pre-diabetic' or 'diabetic' is increasingly seen as artificial. Furthermore, most micro and macrovascular complications may be present already at the pre-diabetic stage.

Hyperglycemia, pre-diabetes and impaired glucose tolerance (IGT) are fully reversible, thus, maintaining normal blood sugar levels is crucial for the prevention and control of diabetes and the various other consequences of the metabolic syndrome. Only interventions that are individually tailored can achieve proper glycemic control, and the glycemic index (GI), which quantifies the glycemic response to particular foods, was developed for this purpose.

In this study the investigators will characterize the blood glucose responses and microbiota of healthy individuals, aiming to assess the influence of food intake on gut microbiota and the influence of gut microbiota on glycemic responses.

DETAILED DESCRIPTION:
Advances in characterization and diagnosis of type 2 Diabetes Mellitus (T2DM) led to the identification of a rapidly growing number of individuals who fall under a 'gray zone' of disturbed yet non-diabetic fasting or post-prandial glucose levels, termed pre-diabetes, impaired glucose tolerance (IGT), or simply individuals with fasting or post-prandial glucose levels in the upper-normal range. All of these poorly characterized groups are at substantial risk for long-term medical complications. Consequently, categorization of glucose levels into 'healthy', 'pre-diabetic' or 'diabetic' is increasingly seen as artificial, and both glucose levels and risk of diabetes are considered as continuous variables. In the past three decades, glucose levels have been rapidly increasing in the overall population in developed and developing countries alike, resulting in a sharp incline in the prevalence of both pre-diabetes and IGT. In the U.S. alone, the estimates are that 79 million people have been affected by 2010, and the projections suggest that 472 million people will be affected worldwide by 2030. Up to 70-90% of those individuals with IGT or pre-diabetes proceed to develop full-blown T2DM. Furthermore, most micro and macrovascular complications, including chronic renal disease, sensory and autonomic neuropathy and diabetic retinopathy, may be present already at the pre-diabetic stage. In addition, pre-diabetic hyperglycemia is linked to multiple manifestations of the metabolic syndrome, such as obesity, hypertension and hypertriglyceridemia, and is an independent risk factor for major macrovascular events such as coronary heart disease and total vascular mortality. Despite these serious risks, and in striking contrast to overt diabetes, hyperglycemia, pre-diabetes and IGT are fully reversible, with up to 55- 80% of individuals reported to revert to normoglycemia and normoinsulinemia upon life-style modifications. Thus, maintaining normal blood sugar levels is crucial for the prevention and control of diabetes and the various other consequences of the metabolic syndrome. The glycemic index (GI), which quantifies the glycemic response to particular foods, was developed for this purpose, but low GI diets have poor predictive value for T2DM development in both the healthy and pre-diabetic settings. This limited success of the GI index may be an inherent problem to any method that assigns a single value to a given food, since individuals vary greatly in their glycemic response to the same food, and even the nature of variation is currently poorly characterized. Along these lines, emerging data from our group and others strongly suggest that proper control and modulation of the glycemic response to foods relies on person-specific factors and thus, only interventions that are individually tailored can achieve proper glycemic control. Although variations in host-related genetic factors affect the normal and post-prandial glycemic response, these factors are estimated to account for only ~10% of the metabolic phenotype. This low estimate is reinforced by the growing incidence of diabetes in recent years. In contrast, increasing importance in glucose homeostasis is being attributed to environmental factors such as the composition and function of the cumulative intestinal microbiota. This immense and poorly understood ecosystem of over 1500 species of bacteria, fungi, and their viruses are modulated by diet, and in turn, profoundly regulate host metabolic processes. Evidence for this host-microbiota interplay includes a distinct microbiota composition found in T2DM patients; and numerous alterations in the microbiome composition and expression of major metabolic pathways found one day after switching from a plant polysaccharide-based diet to a sugary "western" diet in germ-free mice inoculated with a human microbiota. Furthermore, microbiota-induced local gut inflammation was recently linked to a propensity for glucose intolerance, which was reversible upon antibiotic treatment. In this study the investigators will characterize the blood glucose responses and microbiota of healthy individuals, aiming to assess the influence of food intake on gut microbiota and the influence of gut microbiota on glycemic responses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Under 18 years of age
* Mental incompetence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Israeli residents and visitors
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-04-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Blood glucose levels | One week

SECONDARY OUTCOMES:
DNA sequencing of the gut microbiota composition | Before or during the glucose testing week

OTHER OUTCOMES:
Change in postprandial glycemic responses (PPGR) | Four weeks Crossover intervention
  Measured only in newly diagnosed T2DM patients
Change in Fructoseamine | Four weeks Crossover intervention
  Measured only in newly diagnosed T2DM patients
Change in HbA1C | Six months
  Measured only in newly diagnosed T2DM patients

CONTACTS AND LOCATIONS:
Overall Officials: Zamir Halpern, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Gastroenterology Institute, Tel Aviv, Israel

REFERENCES:
- [Derived] Rein M, Ben-Yacov O, Godneva A, Shilo S, Zmora N, Kolobkov D, Cohen-Dolev N, Wolf BC, Kosower N, Lotan-Pompan M, Weinberger A, Halpern Z, Zelber-Sagi S, Elinav E, Segal E. Effects of personalized diets by prediction of glycemic responses on glycemic control and metabolic health in newly diagnosed T2DM: a randomized dietary intervention pilot trial. BMC Med. 2022 Feb 9;20(1):56. doi: 10.1186/s12916-022-02254-y. PMID 35135549
- [Derived] Zeevi D, Korem T, Zmora N, Israeli D, Rothschild D, Weinberger A, Ben-Yacov O, Lador D, Avnit-Sagi T, Lotan-Pompan M, Suez J, Mahdi JA, Matot E, Malka G, Kosower N, Rein M, Zilberman-Schapira G, Dohnalova L, Pevsner-Fischer M, Bikovsky R, Halpern Z, Elinav E, Segal E. Personalized Nutrition by Prediction of Glycemic Responses. Cell. 2015 Nov 19;163(5):1079-1094. doi: 10.1016/j.cell.2015.11.001. PMID 26590418
- [Derived] Korem T, Zeevi D, Suez J, Weinberger A, Avnit-Sagi T, Pompan-Lotan M, Matot E, Jona G, Harmelin A, Cohen N, Sirota-Madi A, Thaiss CA, Pevsner-Fischer M, Sorek R, Xavier R, Elinav E, Segal E. Growth dynamics of gut microbiota in health and disease inferred from single metagenomic samples. Science. 2015 Sep 4;349(6252):1101-1106. doi: 10.1126/science.aac4812. Epub 2015 Jul 30. PMID 26229116